CLINICAL TRIAL: NCT00117260
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a 91-Day Extended-Cycle Combination Oral Contraceptive (Seasonale) for the Treatment of Low Bone Mineral Density in Adolescent Females With Secondary Amenorrhea and Osteopenia
Brief Title: Study to Evaluate the Safety and Efficacy of Seasonale for Treatment of Low Bone Mineral Density
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Research, Inc
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEA-305
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Osteopenia
Keywords: osteopenia; bone mineral density; amenorrhea; adolescents
MeSH Terms: conditions — Bone Diseases, Metabolic; Amenorrhea | interventions — Seasonale; Levonorgestrel; Ethinyl Estradiol

INTERVENTIONS:
Drug: Seasonale (levonorgestrel and ethinyl estradiol)

SUMMARY:
This is a randomized, multicenter, placebo-controlled study to evaluate the effects of Seasonale, an extended-regimen oral contraceptive, on bone mineral density in adolescent females who have had their menstrual period but now have secondary amenorrhea and also have osteopenia. The duration of the study for each patient will be approximately two years.

ELIGIBILITY:
Inclusion Criteria:

* Not sexually active and agree to remain sexually inactive throughout the course of the study
* First menstrual period at least one year ago
* No menstrual period in the last 6 months

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding
* Known or suspected pregnancy
* Medical history of any disorder that contraindicates the use of oral contraceptives

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean percent change in the lumbar spine bone mineral density at month 12

SECONDARY OUTCOMES:
Interim and 24 month mean percent change in lumbar spine bone mineral density
Mean percent change in the proximal femur (hip) bone mineral density
Mean percent change in total body bone mineral density
Mean change in biochemical markers of bone resorption and bone formation
Change in body weight